CLINICAL TRIAL: NCT06307106
Title: Various Strategies to Reduce Acute Post Hemorrhoidectomy Pain: A Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Zakaria Mohamed Ahmed, Principal Investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: #40\14-Jan-2024
Record Dates: First submitted 2024-03-06; First posted 2024-03-12 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-03

CONDITIONS: Acute Post Operative Pain
Keywords: hemorrhoidectomy; acute pain; corticosteroids
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Ketorolac; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- group A: ketorolac and light marcaine injection (Experimental)
  Interventions: Drug: ketorolac and light marcaine
- group B: light marcaine injection (Experimental)
  Interventions: Drug: light marcaine
- group C: corticosteroids injection (Experimental)
  Interventions: Drug: Corticosteroids injection
- group D: topical diclofenac sodium (Experimental)
  Interventions: Drug: Diclofenac Sodium Gel
- control group (Sham Comparator): control group was given the ordinary analgesic protocol without local analgesic application
  Interventions: Other: the standard analgesic protocol

INTERVENTIONS:
Drug: ketorolac and light marcaine — local injection at surgical site of 30 mg ketorolac and 7-1.5 mg\kg\dose light marcaine
  Arms: group A: ketorolac and light marcaine injection
Drug: light marcaine — local injection at surgical site of 7-1.5 mg\kg\dose light marcaine
  Arms: group B: light marcaine injection
Drug: Corticosteroids injection — local injection at surgical site of 40 mg\ dose of dexamethasone
  Arms: group C: corticosteroids injection
Drug: Diclofenac Sodium Gel — topical application of Diclofenac Sodium Gel
  Arms: group D: topical diclofenac sodium
Other: the standard analgesic protocol — the routine analgesia was given without local analgesia application
  Arms: control group

SUMMARY:
Since post hemorrhoidectomy pain is a severe and common post operative symptom so there is a need to find a suitable method for reducing this pain, up to our knowledge, this the first study in ZUH to compare between ketrolac, light Marcaine, corticosteroids and diclofenac sodium injection at surgical site for relieve of post operative pain. This is a randomized controlled comparative prospective clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* both sex.
* age from 18 to 60.

Exclusion Criteria:

* patient refusal.
* patients with associated ano-rectal diseases such as fissures, fistulas, ano-proctitis, recurrent or thrombosed hemorrhoids and ano-rectal malignancy.
* patients with liver cell failure. patients unfit for surgery according to American Society of Anesthesiologists.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2024-01-14 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
age | within 2 days before operation
  adults from 18 to 60 years old
sex | within 2 days before operation
  both sex were included
number of hemorrhoids | within 2 days before operation and intra-operatively
  number of hemorrhoids clinically assessed
degree of hemorroids | within 2 days before operation and intra-operatively
  degree of hemorroids clinically assessed
post operative pain | 1st, 2nd 3rd, 7th, 14th days post-operatively
  post operative assessed using visual analogue scale, minimum score is zero means painless and maximum score 10 means very painful
ambulation | from 1st to 3rd day post-operatively
  early ambulation is evaluated in patients post-operatively
return to work | from one day to one month post-operatively
  first time to return to work is evaluated
patient satisfaction | from one day to one month post-operatively
  patient satisfaction about post-operative pain is assessed using customer satisfaction score. Minimum score is 0 and means very unsatisfied, maximum score is 10 and means very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Reham Zakaria, PhD, Study Chair — faculty of medicine Zagazig University
Locations (1):
- Zagazig University Hospitals, Zagazig, zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No
After completion the study, interested researchers can contact us for providing any data